CLINICAL TRIAL: NCT00616304
Title: Safety and Preliminary Efficacy, Pharmacokinetics, Pharmacodynamics of L-arginine in Severe Falciparum Malaria
Brief Title: Safety and Preliminary Efficacy of L-arginine in Severe Falciparum Malaria
Acronym: ARGISM
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Local circumstances & difficulties in site access has prevented continuation
Sponsor: Menzies School of Health Research (Other)
Collaborators: Wellcome Trust (Other); National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: arginineSM1
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Severe Falciparum Malaria
Keywords: severe falciparum malaria
MeSH Terms: conditions — Malaria, Falciparum | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): L-arginine infusion
  Interventions: Drug: L-arginine hydrochloride
- S (Placebo Comparator): Normal saline infusion
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: L-arginine hydrochloride — Patients will be randomized in two blocks of 18. The first block of 18 patients will receive either 12 g L-arginine or saline placebo. If safety is demonstrated in the first block, a further 18 patients will be enrolled in the second block and randomized to receive either 24g arginine or saline placebo Block 1: Standard RSMM artesunate regimen for severe falciparum malaria plus 12g of L-arginine diluted to a 10% solution and given over 8 hours (n=12); Block 2: Standard RSMM artesunate regimen for severe falciparum malaria plus a 24g dose of L-arginine diluted to a 10% solution given over 8 hours (n=12) Phase 2b: To evaluate any additional benefits of a longer infusion, a further 24 patients will receive L-arginine infusion 1.5g/hour for 24 hours
  Other Names: L-arginine hydrochloride (Pharmalab, Australia)
  Arms: A
Other: Normal saline — Patients with severe malaria will be randomized in two blocks of 18. The first block of 18 patients will receive either 12 g L-arginine or saline placebo. If safety is demonstrated in the first block, a further 18 patients will be enrolled in the second block and randomized to receive either 24g arginine or saline placebo. Blocks 1 and 2: Standard RSMM antimalarial artesunate regimen for severe falciparum malaria plus saline placebo, 240 ml given over 8 hours (n=12).
  Arms: S

SUMMARY:
Background: Mortality from severe malaria remains ~15% despite the use of the most rapidly parasiticidal antimalarial therapy, artesunate. Adjunctive treatments may improve outcome. Our overall goal is to determine if adjunctive treatment with L-arginine is safe and improves outcomes in severe malaria. In studies to date, we have shown that L-arginine is safe in moderately severe malaria, increases nitric oxide production and improves endothelial function. We now propose to extend these studies to patients with severe malaria.

Aims: To determine the safety, preliminary efficacy, pharmacokinetics and pharmacodynamics of L-arginine infusion in severe malaria.

Hypothesis: L-arginine will improve endothelial function, lactate clearance time and tissue oxygen delivery compared to saline with no clinically significant adverse effects.

Methods: Based on previous pharmacokinetic modeling and simulations, we propose a phase 2A randomised controlled trial of L-arginine vs saline in severe malaria, each given over 8 hours. If safety is demonstrated this will be followed by a phase 2B open-label study of 24-hour infusion of L-arginine in severe malaria with safety and preliminary efficacy compared with the 8 hour infusions given in phase 2A.

The primary outcomes will be the improvement in endothelial function and lactate clearance in patients given L-arginine infusion compared with those who received saline. Among the secondary outcomes will be safety and the effect of L-arginine vs saline on tissue oxygen delivery (NIRS).

Data from both phase 2A and 2B will be used to generate a pharmacokinetic/ pharmacodynamic model.

DETAILED DESCRIPTION:
See brief summary

ELIGIBILITY:
Inclusion Criteria:

1. age 18-60 years
2. informed consent obtained
3. time of commencement of artesunate ≤18 hrs before infusion of L-arginine
4. any level of P. falciparum parasitemia, and one or more of the following criteria: i. acute renal failure (creatinine >265umol/L) ii. hyperbilirubinemia (total bilirubin >50 umol/L) with either renal impairment (creatinine >130umol/L) or parasitemia of >100,000 parasites/uL iii. blackwater fever iv. hyperparasitemia (>10% parasitised red cells) v. cerebral malaria (Glasgow coma score <11) vi. Hypoglycemia vii. Respiratory distress (RR >32)

Exclusion Criteria:

1. pregnancy or lactation
2. diabetes
3. serious pre-existing disease (cardiac, hepatic, kidney)
4. systolic blood pressure <90 mmHg after fluid resuscitation
5. initial iSTAT test showing any of the following values: i. K+ > 5.5 meq/L ii. Cl- > 110 meq/L iii. HCO3- < 15 meq/L
6. known allergy to L-arginine
7. evidence of concurrent bacterial infection
8. concurrent therapy with any of the following medications: iv. spironolactone, v. oral nitrates, vi. phosphodiesterase inhibitor (eg sildenafil [Viagra]) vii. alpha-blocking antihypertensive agents (eg prazosin) viii. L-arginine

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2008-02; Primary Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Improvement in endothelial function and lactate clearance. | Endothelial function: end of 8 hour infusion. Lactate clearance: area under the curve until lactate returns to the upper limit of normal

SECONDARY OUTCOMES:
Safety: Clinical and biochemical measures. | During and after infusion. In those receiving L-arginine, biochemical and hemodynamic measures at the completion of infusion will also be compared with measures at the start of infusion.
Change in endothelial function in each arginine infusion regimen vs saline placebo combined | 1 hour response and end of infusion response
Paired change in endothelial function | paired comparison of post-vs pre-infusion values, overall, and in each arginine infusion regimen
Lactate clearance for each infusion regimen | Time for lactate to return to upper limit of normal
Lactate:pyruvate ratio | area under curve/time to normal
Fever clearance time | Fever clearance time
parasite clearance time | parasite clearance time
Change in L-arginine concentration | at 1 and 8 hours
Improvement in microvascular obstruction (OPS) | at 1 and 8 hours
Tissue oxygen consumption and delivery (NIRS) | one and eight hours
change in exhaled NO | one and eight hours
improvement in endothelial activation (decrease in angiopoietin-2 concentrations) | area under curve
improvement in RHPAT among those with baseline dysfunction (RHPAT<1.67) | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas M Anstey, MBBS, Principal Investigator — Menzies School of Health Research; Emiliana Tjitra, MD, Principal Investigator — National Institute of Health Research and Development
Locations (1):
- Mitra Masyarakat Hospital, Timika, Special Region of Papua, Indonesia

REFERENCES:
- [Background] Yeo TW, Lampah DA, Gitawati R, Tjitra E, Kenangalem E, McNeil YR, Darcy CJ, Granger DL, Weinberg JB, Lopansri BK, Price RN, Duffull SB, Celermajer DS, Anstey NM. Impaired nitric oxide bioavailability and L-arginine reversible endothelial dysfunction in adults with falciparum malaria. J Exp Med. 2007 Oct 29;204(11):2693-704. doi: 10.1084/jem.20070819. Epub 2007 Oct 22. PMID 17954570
- [Derived] Yeo TW, Lampah DA, Rooslamiati I, Gitawati R, Tjitra E, Kenangalem E, Price RN, Duffull SB, Anstey NM. A randomized pilot study of L-arginine infusion in severe falciparum malaria: preliminary safety, efficacy and pharmacokinetics. PLoS One. 2013 Jul 29;8(7):e69587. doi: 10.1371/journal.pone.0069587. Print 2013. PMID 23922746